CLINICAL TRIAL: NCT01777724
Title: Evaluation of a Parenting and Stress Management Programme: An Exploratory Randomised Controlled Trial of Triple P-Positive Parenting Program and Stress Control
Brief Title: Evaluation of a Parenting and Stress Management Programmme
Acronym: HAPPY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to time constraints and the withdrawal of Stress Control from the NHS Greater Glasgow and Clyde services.
Sponsor: Medical Research Council (Other Government)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Dr Marion Henderson, Senior Investigator Scientist, Medical Research Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5TK90 HAPPY; U1111-1137-1053 (Other: World Health Organisation Universal Trial Number)
Record Dates: First submitted 2012-12-14; First posted 2013-01-29 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Parenting; Parent Mental Health; Child Behaviour Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention is a combination of Triple P Discussion Groups and Stress Control
  Interventions: Behavioral: Combination of Triple P Discussion Groups and Stress Control
- Control (No Intervention): Waitlist control. Participants allocated to the waitlist control will be able to access the intervention after post-intervention equivalent measures have been completed.

INTERVENTIONS:
Behavioral: Combination of Triple P Discussion Groups and Stress Control — The intervention consists of eight group sessions: two 120 minute Triple P Discussion Group sessions (http://www.triplep.net/), and six 90 minute Stress Control sessions (http://glasgowsteps.com/home.php).
  Arms: Intervention

SUMMARY:
The study will use a randomised controlled trial design to evaluate the effects of a combined intervention of Triple P-Positive Parenting Program Discussion Groups and Stress Control in comparison to a waitlist condition. The combined intervention will be evaluated with parents in Glasgow, United Kingdom, with a 3-8 year old child.

ELIGIBILITY:
Inclusion Criteria:

* Has a child aged between 3 and 8 years old
* Able to attend the group sessions held at Langside Halls, Shawlands in Glasgow, United Kingdom
* Able to read a newspaper without assistance

Exclusion Criteria:

* Child has a diagnosis of a developmental or intellectual disability or other significant health impairment

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in dysfunctional parenting practices as measured by the Parenting Scale | Baseline, mid-intervention (approximately 4 weeks after baseline), post-intervention (approximately 12 weeks after baseline), 3-month follow-up (approximately 24 weeks after baseline)
  Measures dysfunctional parenting practices: laxness, overreactivity, and verbosity
Change in symptoms of depression, anxiety and stress as measured by the Depression Anxiety Stress Scales 21 | Baseline, mid-intervention (approximately 4 weeks after baseline), post-intervention (approximately 12 weeks after baseline), 3-month follow-up (approximately 24 weeks after baseline)

SECONDARY OUTCOMES:
Change in the frequency of disruptive child behaviours as measured by Eyberg Child Behavior Inventory-Intensity scale | Baseline, post-intervention (approximately 12 weeks after baseline), 3-month follow-up (approximately 24 weeks after baseline)
  Measures parents' perceptions of their child's disruptive behaviour
Change in positive mental wellbeing as measured by the Short Warwick-Edinburgh Mental Well-being Scale | Baseline, post-intervention (approximately 12 weeks after baseline), 3-month follow-up (approximately 24 weeks after baseline)
Change in parents' perceptions of their parenting experiences as measured by the Parenting Experience Survey | Baseline, post-intervention (approximately 12 weeks after baseline), 3-month follow-up (approximately 24 weeks after baseline)
Change in parents' perceptions of their parenting self-efficacy as measured by the Child Adjustment and Parent Efficacy Scale-Parent Efficacy subscale | Baseline, post-intervention (approximately 12 weeks after baseline), 3-month follow-up (approximately 24 weeks after baseline)
Change in parents' perceptions of their family relationships as measured by the Parenting and Family Adjustment Scale-Family Relationships subscale | Baseline, post-intervention (approximately 12 weeks after baseline), 3-month follow-up (approximately 24 weeks after baseline)

OTHER OUTCOMES:
Family demographics | Baseline
  Demographic information of the participating families
Parents' satisfaction with the Triple P Discussion Groups and Stress Control, as measured by the Consumer Satisfaction Questionnaire developed for Triple P programmes, and the Consumer Satisfaction Questionnaire developed for Stress Control | Post-intervention (approximately 12 weeks after baseline)
The fidelity of the intervention as measured by the Triple P Discussion Group session content checklists, and session content checklists for Stress Control that were developed for this study | The practitioner/s delivering the intervention will complete a session content checklist after each Triple P Discussion Group and after each Stress Control session

CONTACTS AND LOCATIONS:
Overall Officials: Marion Henderson, PhD, Principal Investigator — Medical Research Council Social and Public Health Sciences Unit
Locations (1):
- Medical Research Council Social and Public Health Sciences Unit, Glasgow, United Kingdom

REFERENCES:
- [Derived] Palmer ML, Henderson M, Sanders MR, Keown LJ, White J. Study protocol: evaluation of a parenting and stress management programme: a randomised controlled trial of Triple P Discussion Groups and Stress Control. BMC Public Health. 2013 Sep 25;13:888. doi: 10.1186/1471-2458-13-888. PMID 24066966
- See also: Medical Research Council Social and Public Health Sciences Unit homepage — http://www.sphsu.mrc.ac.uk/